CLINICAL TRIAL: NCT06992453
Title: Disentangling Microbiome Engraftment by Multi-omics of the Gut Ecosystem During Fecal Transplant
Brief Title: Multi-omics Dissection of Gut Microbiome Engraftment During FMT
Acronym: DissEcT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Gianluca Ianiro, Principal Investigator, MD, PhD, Catholic University of the Sacred Heart
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 7416
Record Dates: First submitted 2025-05-13; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Recurrent C. Difficile (rCDI); Ulcerative Colitis (UC); Metabolic Syndrome (MetS)
Keywords: Microbiome engraftment; Gut ecosystem; Fecal microbiota transplantation
MeSH Terms: conditions — Colitis, Ulcerative; Metabolic Syndrome | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Recurrent C. difficile infection (rCDI) Cohort (Experimental): Patients with recurrent C. difficile infection (rCDI) will be recruited among those referred to the Digestive Disease Centre (CEMAD) of the Fondazione Policlinico Universitario A. Gemelli IRCCS. Patients with all inclusion criteria and none of the exclusion criteria will be considered for this study.
  Interventions: Other: Fecal microbiota transplantation (FMT)
- Ulcerative Colitis (UC) Cohort (Experimental): Patients with Ulcerative Colitis (UC) will be recruited among those referred to the Digestive Disease Centre (CEMAD) of the Fondazione Policlinico Universitario A. Gemelli IRCCS. Patients with all inclusion criteria and none of the exclusion criteria will be considered for this study.
  Interventions: Other: Fecal microbiota transplantation (FMT)
- Metabolic syndrome (MetS) Cohort (Experimental): Patients with metabolic syndrome (MetS), will be recruited among those referred to the Digestive Disease Centre (CEMAD) and to the Endocrine and Metabolic Diseases Unit of the Fondazione Policlinico Universitario A. Gemelli IRCCS.
  Interventions: Other: Fecal microbiota transplantation (FMT)

INTERVENTIONS:
Other: Fecal microbiota transplantation (FMT) — Patients will receive a first donor FMT by colonoscopy, after a pre-conditioning with vancomycin and neomycin + bacitracin for 3 days, because data from our group show that pre-FMT antibiotics are associated with higher rates of microbial engraftment. Then they will receive two cycles, respectively after 3 and 7 days after colonoscopy - FMT, of frozen donor FMT capsules (15 capsules b.i.d. per 3 days). Patients will always receive feces from the same donor.

SUMMARY:
The gut microbiota plays a key role in immunity and metabolism and contributes to diseases such as recurrent C. difficile infection (rCDI), ulcerative colitis (UC), and metabolic syndrome (MetS). Microbiota therapeutics, particularly fecal microbiota transplantation (FMT), show promise-achieving ~90% cure rates in rCDI-but demonstrate variable efficacy in chronic conditions. Microbiome engraftment appears critical for FMT success, yet consistent predictors remain lacking. A meta-analysis of 20 FMT studies by our group and the Segata Lab linked engraftment to clinical response across diseases, with taxon-specific patterns and ML-based predictability. While viral, fungal, host immune, genetic, and metabolic factors may affect engraftment, their roles are not well-defined. Key unresolved questions include the interplay among host factors, microbial strains, and metabolites, their influence on engraftment, and impact on clinical outcomes. This study aims to unravel microbiome engraftment dynamics and link them to therapeutic response.

DETAILED DESCRIPTION:
Gut microbiota regulates key functions in humans, i.e. immunity and metabolism, and is a pathogenic pathway of many disorders, including recurrent C. difficile infection (rCDI), ulcerative colitis (UC), and metabolic syndrome (MetS). Microbiota therapeutics (MT) have raised high expectations without comparable results. Among MT, fecal microbiota transplantation (FMT), the transfer of healthy donor feces to a recipient with a microbiome-associated disease, has achieved high (nearly 90%) cure rates of rCDI but lower and less consistent results in chronic disorders, i.e. UC or MetS. Clinical and microbial features seem to be related with FMT outcomes, but consistent predictors are not available.

Donor-recipient microbiome engraftment may be critical for the clinical success of FMT. In a pooled meta-analysis of 20 FMT studies in different diseases by our group and the Segata Lab , donor recipient microbiome engraftment was associated with clinical response regardless of disease, differed among bacterial taxa, and was predicted by machine learning (ML). Other factors could influence engraftment, but evidence is unclear. Virome and fungome, have been linked to FMT success, but their engraftment kinetics is unknown. Host factors, i.e. genetics, gut immunity and microbial metabolites are supposed to play a role in engraftment, but supporting data are still absent.

Crucial issues of the engraftment dynamics remain still unsolved, including 1) which are the interactions among host factors, microbial strains, and products during FMT; 2)whether and how they influence engraftment and 3) clinical outcomes.Our aim is to disentangle the dynamics of microbiome engraftment and correlate them to clinical outcomes.

OBJECTIVES

Primary objectives - To assess the longitudinal multidomain interactions of host and microbiome variables and their influence on microbial engraftment

Secondary Objectives

- To assess the longitudinal multidomain interactions of host and microbiome variables and their influence on clinical outcomes

Endpoints

Primary - The longitudinal evaluation of multidomain interactions of host and microbiome variables throughout a multi-omics approach at 90 days after the last FMT

Secondary

- The longitudinal evaluation of multidomain interactions of host and microbiome variables throughout a multi-omics approach at 7,30,180,360 days after the last FMT

Procedures:

Baseline assessment

At baseline enrolled patients will be evaluated by the gastroenterology staff and endocrine and metabolic Unit staff of the Fondazione Policlinico Universitario A. Gemelli IRCCS and their demographic, clinical characteristics and laboratory data will be recorded, specifically:

* Disease clinical and endoscopic activity for UC patients, expressed using Mayo score
* Insulin sensitivity, assessed by Matsuda index and OGIS index after an oral glucose tolerance test (OGTT), for MetS patients.
* Clinical characteristic, the occurrence of diarrhea and fecal C. difficile toxin, in patients affected by recurrent CDI

In addition, the following data for patients in all cohorts will be collected:

* Erythrocyte Sedimentation Rate (ESR) and C Reactive Protein (CRP) serum levels.
* White Blood Count, Red Blood Count, serum creatinine, aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma-glutamyl transferase (GGT), urine analysis. At baseline (pre - FMT), a blood and stool sample, and gut (colonic) biopsy will be collected.

After the baseline assessment, all patients will undergo to the FMT combined (colonoscopy + capsules) procedure.

Follow-up visits

All patients will undergo follow-up visits at day 7, 30, 60, 90, 180, 360 after the last FMT.

At each time point, the gastroenterology staff and endocrine and metabolic unit staff of the Fondazione Policlinico Universitario A. Gemelli IRCCS, will assess the same items assessed at baseline (demographic, clinical characteristics including disease activity, and laboratory data) and the same blood and stool sample will be collected. Moreover, a stool sample will be collected after the pre-conditioning with nonabsorbable antibiotics.

Gut biopsies will be collected at day 30, 90, 180 and 360 after the last FMT.

Treatment

Patients will receive a first donor FMT by colonoscopy, after a pre-conditioning with vancomycin and neomycin + bacitracin for 3 days, because data from our group show that pre-FMT antibiotics are associated with higher rates of microbial engraftment. Then they will receive two cycles, respectively after 3 and 7 days after colonoscopy - FMT, of frozen donor FMT capsules (15 capsules b.i.d. per 3 days). Patients will always receive feces from the same donor.

Donors Recruitment

Potential donor candidates will be evaluated by the gastroenterology staff of the Fondazione Policlinico Universitario A. Gemelli IRCCS, following protocols recommended by international guidelines and according to the recent recommendations imposed by the reorganization of faecal microbiota transplant during the COVID-19 pandemic.

In addition, in relation to the national and international spread of human cases of monkey pox, according to the reports of the European Centre for Disease Prevention and Control (ECDC) and the FDA and as indicated in the circulars of the General Directorate for Health Prevention of the National Ministry of Health of 25/5/2022 (Prot. DGPREV 0026837), of 02/08/2022 (Prot. DGPREV 0034905) and in The National Transplants Center note of 07/06/2022 (Prot. ISS 0021745).

Collection and storage of stool and blood samples

Stool samples will be collected in donors and in patients at baseline and at each follow-up visit, using a Zymo buffer, to preserve feces at room temperature for up to 48 hours. Fecal samples will be stored at -80°C and assigned de-identified IDs. Blood samples will be collected in donors and in patients at each timepoint (1 mL of whole blood per sample), centrifuged at 2000 rpm for 15 minutes for serum collection, stored at a temperature of -80°C. Both stool and blood samples will be stored until the end of the clinical study (after the end of the follow-up of the last enrolled patient). Then, blood samples will be used for the analysis of human genes, associated with microbiome and beta diversity, while stool samples will be used for microbiome analysis.

RNA extraction

Total RNA will be prepared by the RNeasy kit (Qiagen) based on manufacturer's instructions. Samples are first lysed and then homogenized. Ethanol is added to the lysate to provide ideal binding conditions. The lysate is then loaded onto the RNeasy silica membrane and RNA binds to the silica membrane, and all contaminants are efficiently washed away. 100 ng/μl of RNA will be analyzed for RNA integrity and then interrogated by microarray using Affymetrix technology. Fold-change data will be calculated for each gene from the microarray analysis, comparing expression among different groups of samples. Data set will be trimmed to include only those genes showing at least a ±1.5-fold change relative to the C. difficile infection cohort, which will be then submitted to Ingenuity Pathway Analysis (IPA, Qiagen) for unsupervised clustering analysis. Potential gene networks will be identified by the Global Molecular Network algorithm.

Genome extraction and shotgun metagenomic sequencing

DNA extraction will be performed by using the Dneasy PowerSoil Pro Kit (QIAGEN, Germany) according to the manufacturer's procedures. DNA concentration will be measured with Qubit (Thermo Fisher Scientific, USA), and DNA will be then stored at - 20°C. Sequencing libraries will be prepared using the Illumina® DNA Prep (M) Tagmentation kit (Illumina, California, USA) following the manufacturer's guidelines.

Shotgun metagenomic sequencing will be performed on the Illumina NovaSeq platform.

A >7.5Gb/sample of 150nt paired end reads (insert size ~150nt) will be generate. This will be sufficient to cover at 2x a 4Mb bacterial, fungal, and viral genome present at an abundance of 0.1% after accounting for human DNA reads removal, and to detect with our markerbased strategy organisms at abundances as low as 0.01%. All the above procedures have been extensively validated. As gut mycobiome is hardly detected by WGS, it will be assessed also by sequencing the ITS2 region and the 18SrRNA gene.

Metagenome quality control and pre-processing

Newly generated shotgun metagenomic sequences will be pre-processed and quality controlled using the pipeline available at https://github.com/SegataLab/preprocessing.

Reads will be quality-controlled and those of low quality (quality score 2 ambiguous nucleotides were removed with Trim Galore. Contaminant and host DNA will be identified with Bowtie2 using the parameter -sensitive-local, allowing confident removal of the phiX 174 Illumina spike-in and human reads (hg19 human genome release). Remaining high-quality reads will be sorted and split to create forward reverse and unpaired reads output files for each metagenome.

Microbiome taxonomic profiling

Microbiome taxonomic profiling will be performed following the general guidelines and relying on the bioBakery computational environment. The taxonomic profiling and quantification of organisms' relative abundances of all metagenomic samples will be quantified using MetaPhlAn 3.0 (species-level profiling) and StrainPhlAn 3 (strain-level profiling).

Metatranscriptomic, metabolomic and metaproteomic analysis

Metatranscriptomics (MTR), metabolomics (MTB) and metaproteomics (MTP) will be performed in stool samples. For a metatrascriptomic analysis sample preparation will use the most up-to-date and validated protocol for mRNA fraction enrichment by rRNA depletion as per the Illumina protocols. cDNA libraries will be synthetized, and dedicated pipelines will follow.

Furthermore, volatile, and nonvolatile metabolites will be assessed in stool samples to perform a metabolomic analysis. The untargeted analysis will be carried out by GC-MS coupled to solid phase microextraction (SPME) (Agilent Technologies 7890B GC, coupled to a 5977A mass selective detector), 1H-NMR (50), and by LC-MS/MS based technology by pipelines optimized in house. Data will be analyzed with MetaboAnalyst, SCIEX OS, MATLAB toolbox, and R and Phyton scripts. Metaproteomics required a specific procedure as follow, microbial cells will be purified from 300 mg of each stool sample and cells lysis will be performed adding 4% SDS (w/v) lysis buffer followed by incubation at 95 °C for 10 min with agitation and 3 rounds of sonication. After protein quantification, equal amount of each sample will be trypsin digested by FASP protocol. The tryptic peptide mixtures will be analyzed by nanoLCESI-MS/MS acquisition on a high resolution mass spectrometer. Data will be analyzed with MetaLab platform and ad-hoc Python scripts.

Cytokine Multiplex Immunoassay

Through Multiplex Bead analysis for the assessment of specific cytokine in biopsy samples will be perform, following manufacturer's instructions. IL-1b, IL-1Ra, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-9, IL-10, IL-12, IL-13, IL-15, IL-17, Eotaxin, FGF basic, G-CSF, GM-CSF, IFN-g, IP-10, MCP-1, MIP-1a, PDGF-bb, MIP-1b, RANTES, TNF-a, VEGF will be analyzed. Flow cytometry will be also performed in colonic biopsies to identify the specific phenotype of immune cells localized in the mucosal samples.

Machine learning analysis

Machine learning models will be used to identify and reproducibly characterize responder and non-responder profiles. In a Python 3.9 environment using scikit-learn (ver. 0.22.1), two unsupervised ML algorithm, K-means and Agglomerative Hierarchical Clustering, will be used for creating patient clusters based on baseline microbiome, cytokine signature and clinical features, in order to assess whether ML may identify distinct subgroups of microbiome and cytokine profiles associated with clinical response.

Statistical Analysis

Sample size calculation

This study is exploratory in nature and sample size calculation is no hypotheses-driven. A size of 30 patients in each group (total sample size 3*30=90 patients) will be considered. As a general approach 30 patients will have an 80% power of detecting large effect size (f=0.40) at a significance level of 5%.

Data Analysis

Descriptive statistics will be used to analyse baseline and follow-up variables.

Data will be presented as mean and standard deviation (SD) or as median and first and third quartile according to the normality of data distribution. Qualitative variables will be summarized by absolute and relative frequencies (percentage). All statistics will be tabulated according to groups (UC, rCDI, MetS) and to different timepoints. According to the data distribution an approach based on analysis of variance or Kruskal-Wallis/Friedmann test will be employed. Due to the high number of variables resulting from analyses and to the exploratory nature of this project no adjustment for multiple testing will be considered. Machine-Learning algorithms will deal with the complexity of the multidimensional data matrix.

SAFETY REPORTING

No specific serious adverse events are expected. Adverse events are defined as any undesirable experience occurring to a subject during the study, whether or not considered related to the surveillance protocol. All adverse events reported spontaneously by the subject or observed by the investigator or his staff will be recorded and reported to the coordinating investigator.

A serious adverse event is any untoward medical occurrence or effect that at any dose:

* results in death;
* is life threatening (at the time of the event);
* requires hospitalization or prolongation of existing inpatients' hospitalization;
* results in persistent or significant disability or incapacity;
* is a congenital anomaly or birth defect;
* is a new event of the trial likely to affect the safety of the subjects, such as an unexpected outcome of an adverse reaction, lack of efficacy of an IMP used for the treatment of a life-threatening disease, major safety finding from a newly completed animal study, etc. All SAEs will be reported by the coordinating investigator to the ethics committee of Fondazione Policlinico "A. Gemelli" IRCCS and to the Italian National Transplant Centre SAEs that result in death or are life threatening should be reported expedited. The expedited reporting will occur not later than 7 days after the responsible investigator has first knowledge of the adverse reaction. This is for a preliminary report with another 8 days for completion of the report. All adverse events will be followed until they have abated or until a stable situation has been reached. Depending on the event, follow up may require additional tests or medical procedures as indicated, and/or referral to the general physician or a medical specialist.

ETHICS

The study protocol must be approved by the ethics committee CET Lazio Area 3 and by the Italian National Transplant Centre will be registered at ClinicalTrials.gov. The study will be conducted in accordance with the Consolidated Standards of Reporting Trials (CONSORT) Statement.

ELIGIBILITY:
Inclusion Criteria:

Coorte: Patients affected by Ulcerative Colitis

* Age ≥18 years.
* Biologic-naïve active UC
* UC with mild-to-moderate activity (total Mayo score 3-10 + endoscopic subscore≥1) (23)
* UC during stable maintenance therapy (> 8 weeks with salicylates, immunosuppressants);
* Ability to give informed consent.

Coorte: Patients affected by metabolic syndrome

* Age ≥18 years.
* Patients with MetS (high glycaemia levels (> 100 mg/dL), hypertension (> 130/85 mmHg), raised triglyceride levels (> 150 mg/dL), low high-density lipoprotein cholesterol levels (< 40 mg/dL in men; <50 mg/dL in women), and abdominal obesity (waist circumference of > 102 cm in men; >88 cm in women)
* Stable treatment (> 8 weeks) of one of these disorders, included in MetS definition.
* Family history of diabetes mellitus type 2
* Polycystic ovary syndrome (PCOs)
* Ability to give informed consent

Coorte: Patients affected by rCDI

* Age ≥18 years
* Mild recurrent Clostridioides difficile infection (26)
* Ability to give informed consent.

Exclusion criteria

* Pregnancy, breastfeeding, and the refusal to follow an effective contraception method for all the study duration (for women).
* Known active gastrointestinal disorders (e.g. infectious gastroenteritis except CDI, coeliac disease, irritable bowel syndrome, chronic pancreatitis, biliary salt diarrhoea) apart from UC, with clinical characteristics reports in inclusion criteria.
* Antimicrobial treatment or use of probiotics up to 4 weeks prior to screening visit (apart for patients with rCDI)
* Previous colorectal surgery or cutaneous stoma
* Critical and severe comorbidities
* Inability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2029-01-19 (Estimated); Study Completion 2029-02-19 (Estimated)

PRIMARY OUTCOMES:
Longitudinal Analysis of Host-Microbiome Interactions Driving Microbial Engraftment | 60 months
  To assess the longitudinal multidomain interactions of host and microbiome variables and their influence on microbial engraftment. Microbiome taxonomic profiling will be performed following the general guidelines and relying on the bioBakery computational environment. The taxonomic profiling and quantification of organisms' relative abundances of all metagenomic samples will be quantified using MetaPhlAn 3.0 (species-level profiling) and StrainPhlAn 3 (strain-level profiling). Metatranscriptomics (MTR), metabolomics (MTB) and metaproteomics (MTP) will be performed in stool samples. Through Multiplex Bead analysis for the assessment of specific cytokine in biopsy samples will be perform, following manufacturer's instructions. Flow cytometry will be also performed in colonic biopsies to identify the specific phenotype of immune cells localized in the mucosal samples.

SECONDARY OUTCOMES:
Longitudinal Analysis of Host-Microbiome Interactions and Their Impact on Clinical Outcomes | 60 months
  A longitudinal multidomain analysis will investigate host-microbiome interactions using taxonomic profiling, metatranscriptomics, metabolomics, and metaproteomics in stool samples. Cytokine profiling in biopsy samples will be performed via Multiplex Bead analysis. These variables will be correlated with clinical outcomes, including disease activity in UC patients (Mayo score), insulin sensitivity in MetS patients (Matsuda and OGIS indices post-OGTT), and clinical features such as diarrhea and fecal C. difficile toxin in recurrent CDI cases.

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of the Sacred Heart, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be shared upon reasonable request for academic research purposes, following approval of a data access proposal and signing of a data use agreement.
Supporting Information: Study Protocol, SAP, ICF
Access Criteria: Data will be given upon reasonable request to the PI.

REFERENCES:
- [Result] D'Haens GR, Jobin C. Fecal Microbial Transplantation for Diseases Beyond Recurrent Clostridium Difficile Infection. Gastroenterology. 2019 Sep;157(3):624-636. doi: 10.1053/j.gastro.2019.04.053. Epub 2019 Jun 17. PMID 31220424
- [Result] Ianiro G, Bibbo S, Gasbarrini A, Cammarota G. Therapeutic modulation of gut microbiota: current clinical applications and future perspectives. Curr Drug Targets. 2014;15(8):762-70. doi: 10.2174/1389450115666140606111402. PMID 24909808
- [Result] Tixier EN, Verheyen E, Luo Y, Grinspan LT, Du CH, Ungaro RC, Walsh S, Grinspan AM. Systematic Review with Meta-Analysis: Fecal Microbiota Transplantation for Severe or Fulminant Clostridioides difficile. Dig Dis Sci. 2022 Mar;67(3):978-988. doi: 10.1007/s10620-021-06908-4. Epub 2021 Mar 22. PMID 33748913
- [Result] Baunwall SMD, Lee MM, Eriksen MK, Mullish BH, Marchesi JR, Dahlerup JF, Hvas CL. Faecal microbiota transplantation for recurrent Clostridioides difficile infection: An updated systematic review and meta-analysis. EClinicalMedicine. 2020 Nov 23;29-30:100642. doi: 10.1016/j.eclinm.2020.100642. eCollection 2020 Dec. PMID 33437951
- [Result] Ianiro G, Eusebi LH, Black CJ, Gasbarrini A, Cammarota G, Ford AC. Systematic review with meta-analysis: efficacy of faecal microbiota transplantation for the treatment of irritable bowel syndrome. Aliment Pharmacol Ther. 2019 Aug;50(3):240-248. doi: 10.1111/apt.15330. Epub 2019 May 28. PMID 31136009
- [Result] Costello SP, Soo W, Bryant RV, Jairath V, Hart AL, Andrews JM. Systematic review with meta-analysis: faecal microbiota transplantation for the induction of remission for active ulcerative colitis. Aliment Pharmacol Ther. 2017 Aug;46(3):213-224. doi: 10.1111/apt.14173. Epub 2017 Jun 14. PMID 28612983
- [Result] Proenca IM, Allegretti JR, Bernardo WM, de Moura DTH, Ponte Neto AM, Matsubayashi CO, Flor MM, Kotinda APST, de Moura EGH. Fecal microbiota transplantation improves metabolic syndrome parameters: systematic review with meta-analysis based on randomized clinical trials. Nutr Res. 2020 Nov;83:1-14. doi: 10.1016/j.nutres.2020.06.018. Epub 2020 Jul 3. PMID 32987284
- [Result] Ianiro G, Sanguinetti M, Gasbarrini A, Cammarota G. Predictors of failure after single faecal microbiota transplantation in patients with recurrent Clostridium difficile infection: results from a 3-year cohort study: authors' reply. Clin Microbiol Infect. 2017 Nov;23(11):891. doi: 10.1016/j.cmi.2017.05.005. Epub 2017 May 11. No abstract available. PMID 28502839
- [Result] Moayyedi P, Surette MG, Kim PT, Libertucci J, Wolfe M, Onischi C, Armstrong D, Marshall JK, Kassam Z, Reinisch W, Lee CH. Fecal Microbiota Transplantation Induces Remission in Patients With Active Ulcerative Colitis in a Randomized Controlled Trial. Gastroenterology. 2015 Jul;149(1):102-109.e6. doi: 10.1053/j.gastro.2015.04.001. Epub 2015 Apr 7. PMID 25857665
- [Result] Ianiro G, Maida M, Burisch J, Simonelli C, Hold G, Ventimiglia M, Gasbarrini A, Cammarota G. Efficacy of different faecal microbiota transplantation protocols for Clostridium difficile infection: A systematic review and meta-analysis. United European Gastroenterol J. 2018 Oct;6(8):1232-1244. doi: 10.1177/2050640618780762. Epub 2018 Jun 3. PMID 30288286
- [Result] Zuo T, Wong SH, Lam K, Lui R, Cheung K, Tang W, Ching JYL, Chan PKS, Chan MCW, Wu JCY, Chan FKL, Yu J, Sung JJY, Ng SC. Bacteriophage transfer during faecal microbiota transplantation in Clostridium difficile infection is associated with treatment outcome. Gut. 2018 Apr;67(4):634-643. doi: 10.1136/gutjnl-2017-313952. Epub 2017 May 24. PMID 28539351
- [Result] Zuo T, Wong SH, Cheung CP, Lam K, Lui R, Cheung K, Zhang F, Tang W, Ching JYL, Wu JCY, Chan PKS, Sung JJY, Yu J, Chan FKL, Ng SC. Gut fungal dysbiosis correlates with reduced efficacy of fecal microbiota transplantation in Clostridium difficile infection. Nat Commun. 2018 Sep 10;9(1):3663. doi: 10.1038/s41467-018-06103-6. PMID 30202057
- [Result] Kootte RS, Levin E, Salojarvi J, Smits LP, Hartstra AV, Udayappan SD, Hermes G, Bouter KE, Koopen AM, Holst JJ, Knop FK, Blaak EE, Zhao J, Smidt H, Harms AC, Hankemeijer T, Bergman JJGHM, Romijn HA, Schaap FG, Olde Damink SWM, Ackermans MT, Dallinga-Thie GM, Zoetendal E, de Vos WM, Serlie MJ, Stroes ESG, Groen AK, Nieuwdorp M. Improvement of Insulin Sensitivity after Lean Donor Feces in Metabolic Syndrome Is Driven by Baseline Intestinal Microbiota Composition. Cell Metab. 2017 Oct 3;26(4):611-619.e6. doi: 10.1016/j.cmet.2017.09.008. PMID 28978426
- [Result] Vaughn BP, Vatanen T, Allegretti JR, Bai A, Xavier RJ, Korzenik J, Gevers D, Ting A, Robson SC, Moss AC. Increased Intestinal Microbial Diversity Following Fecal Microbiota Transplant for Active Crohn's Disease. Inflamm Bowel Dis. 2016 Sep;22(9):2182-90. doi: 10.1097/MIB.0000000000000893. PMID 27542133
- [Result] Turpin W, Espin-Garcia O, Xu W, Silverberg MS, Kevans D, Smith MI, Guttman DS, Griffiths A, Panaccione R, Otley A, Xu L, Shestopaloff K, Moreno-Hagelsieb G; GEM Project Research Consortium; Paterson AD, Croitoru K. Association of host genome with intestinal microbial composition in a large healthy cohort. Nat Genet. 2016 Nov;48(11):1413-1417. doi: 10.1038/ng.3693. Epub 2016 Oct 3. PMID 27694960
- [Result] Goodrich JK, Davenport ER, Clark AG, Ley RE. The Relationship Between the Human Genome and Microbiome Comes into View. Annu Rev Genet. 2017 Nov 27;51:413-433. doi: 10.1146/annurev-genet-110711-155532. Epub 2017 Sep 20. PMID 28934590
- [Result] Danne C, Rolhion N, Sokol H. Recipient factors in faecal microbiota transplantation: one stool does not fit all. Nat Rev Gastroenterol Hepatol. 2021 Jul;18(7):503-513. doi: 10.1038/s41575-021-00441-5. Epub 2021 Apr 27. PMID 33907321
- [Result] Littmann ER, Lee JJ, Denny JE, Alam Z, Maslanka JR, Zarin I, Matsuda R, Carter RA, Susac B, Saffern MS, Fett B, Mattei LM, Bittinger K, Abt MC. Host immunity modulates the efficacy of microbiota transplantation for treatment of Clostridioides difficile infection. Nat Commun. 2021 Feb 2;12(1):755. doi: 10.1038/s41467-020-20793-x. PMID 33531483
- [Result] Lewis JD, Chuai S, Nessel L, Lichtenstein GR, Aberra FN, Ellenberg JH. Use of the noninvasive components of the Mayo score to assess clinical response in ulcerative colitis. Inflamm Bowel Dis. 2008 Dec;14(12):1660-6. doi: 10.1002/ibd.20520. PMID 18623174
- [Result] Lavelle A, Sokol H. Gut microbiota-derived metabolites as key actors in inflammatory bowel disease. Nat Rev Gastroenterol Hepatol. 2020 Apr;17(4):223-237. doi: 10.1038/s41575-019-0258-z. Epub 2020 Feb 19. PMID 32076145
- [Result] Khoruts A, Sadowsky MJ. Understanding the mechanisms of faecal microbiota transplantation. Nat Rev Gastroenterol Hepatol. 2016 Sep;13(9):508-16. doi: 10.1038/nrgastro.2016.98. Epub 2016 Jun 22. PMID 27329806
- [Result] Zimmet P, Magliano D, Matsuzawa Y, Alberti G, Shaw J. The metabolic syndrome: a global public health problem and a new definition. J Atheroscler Thromb. 2005;12(6):295-300. doi: 10.5551/jat.12.295. PMID 16394610
- [Result] Alberti KG, Eckel RH, Grundy SM, Zimmet PZ, Cleeman JI, Donato KA, Fruchart JC, James WP, Loria CM, Smith SC Jr; International Diabetes Federation Task Force on Epidemiology and Prevention; Hational Heart, Lung, and Blood Institute; American Heart Association; World Heart Federation; International Atherosclerosis Society; International Association for the Study of Obesity. Harmonizing the metabolic syndrome: a joint interim statement of the International Diabetes Federation Task Force on Epidemiology and Prevention; National Heart, Lung, and Blood Institute; American Heart Association; World Heart Federation; International Atherosclerosis Society; and International Association for the Study of Obesity. Circulation. 2009 Oct 20;120(16):1640-5. doi: 10.1161/CIRCULATIONAHA.109.192644. Epub 2009 Oct 5. PMID 19805654
- [Result] McDonald LC, Gerding DN, Johnson S, Bakken JS, Carroll KC, Coffin SE, Dubberke ER, Garey KW, Gould CV, Kelly C, Loo V, Shaklee Sammons J, Sandora TJ, Wilcox MH. Clinical Practice Guidelines for Clostridium difficile Infection in Adults and Children: 2017 Update by the Infectious Diseases Society of America (IDSA) and Society for Healthcare Epidemiology of America (SHEA). Clin Infect Dis. 2018 Mar 19;66(7):987-994. doi: 10.1093/cid/ciy149. PMID 29562266
- [Result] Costello SP, Hughes PA, Waters O, Bryant RV, Vincent AD, Blatchford P, Katsikeros R, Makanyanga J, Campaniello MA, Mavrangelos C, Rosewarne CP, Bickley C, Peters C, Schoeman MN, Conlon MA, Roberts-Thomson IC, Andrews JM. Effect of Fecal Microbiota Transplantation on 8-Week Remission in Patients With Ulcerative Colitis: A Randomized Clinical Trial. JAMA. 2019 Jan 15;321(2):156-164. doi: 10.1001/jama.2018.20046. PMID 30644982
- [Result] Matsuda M, DeFronzo RA. Insulin sensitivity indices obtained from oral glucose tolerance testing: comparison with the euglycemic insulin clamp. Diabetes Care. 1999 Sep;22(9):1462-70. doi: 10.2337/diacare.22.9.1462. PMID 10480510
- [Result] Mari A, Pacini G, Murphy E, Ludvik B, Nolan JJ. A model-based method for assessing insulin sensitivity from the oral glucose tolerance test. Diabetes Care. 2001 Mar;24(3):539-48. doi: 10.2337/diacare.24.3.539. PMID 11289482
- [Result] Cammarota G, Masucci L, Ianiro G, Bibbo S, Dinoi G, Costamagna G, Sanguinetti M, Gasbarrini A. Randomised clinical trial: faecal microbiota transplantation by colonoscopy vs. vancomycin for the treatment of recurrent Clostridium difficile infection. Aliment Pharmacol Ther. 2015 May;41(9):835-43. doi: 10.1111/apt.13144. Epub 2015 Mar 1. PMID 25728808
- [Result] Baruch EN, Youngster I, Ben-Betzalel G, Ortenberg R, Lahat A, Katz L, Adler K, Dick-Necula D, Raskin S, Bloch N, Rotin D, Anafi L, Avivi C, Melnichenko J, Steinberg-Silman Y, Mamtani R, Harati H, Asher N, Shapira-Frommer R, Brosh-Nissimov T, Eshet Y, Ben-Simon S, Ziv O, Khan MAW, Amit M, Ajami NJ, Barshack I, Schachter J, Wargo JA, Koren O, Markel G, Boursi B. Fecal microbiota transplant promotes response in immunotherapy-refractory melanoma patients. Science. 2021 Feb 5;371(6529):602-609. doi: 10.1126/science.abb5920. Epub 2020 Dec 10. PMID 33303685
- [Result] Cammarota G, Ianiro G, Kelly CR, Mullish BH, Allegretti JR, Kassam Z, Putignani L, Fischer M, Keller JJ, Costello SP, Sokol H, Kump P, Satokari R, Kahn SA, Kao D, Arkkila P, Kuijper EJ, Vehreschild MJG, Pintus C, Lopetuso L, Masucci L, Scaldaferri F, Terveer EM, Nieuwdorp M, Lopez-Sanroman A, Kupcinskas J, Hart A, Tilg H, Gasbarrini A. International consensus conference on stool banking for faecal microbiota transplantation in clinical practice. Gut. 2019 Dec;68(12):2111-2121. doi: 10.1136/gutjnl-2019-319548. Epub 2019 Sep 28. PMID 31563878
- [Result] Ianiro G, Mullish BH, Kelly CR, Kassam Z, Kuijper EJ, Ng SC, Iqbal TH, Allegretti JR, Bibbo S, Sokol H, Zhang F, Fischer M, Costello SP, Keller JJ, Masucci L, van Prehn J, Quaranta G, Quraishi MN, Segal J, Kao D, Satokari R, Sanguinetti M, Tilg H, Gasbarrini A, Cammarota G. Reorganisation of faecal microbiota transplant services during the COVID-19 pandemic. Gut. 2020 Sep;69(9):1555-1563. doi: 10.1136/gutjnl-2020-321829. Epub 2020 Jul 3. PMID 32620549
- [Result] El-Salhy M, Hatlebakk JG, Gilja OH, Brathen Kristoffersen A, Hausken T. Efficacy of faecal microbiota transplantation for patients with irritable bowel syndrome in a randomised, double-blind, placebo-controlled study. Gut. 2020 May;69(5):859-867. doi: 10.1136/gutjnl-2019-319630. Epub 2019 Dec 18. PMID 31852769
- [Result] Youngster I, Mahabamunuge J, Systrom HK, Sauk J, Khalili H, Levin J, Kaplan JL, Hohmann EL. Oral, frozen fecal microbiota transplant (FMT) capsules for recurrent Clostridium difficile infection. BMC Med. 2016 Sep 9;14(1):134. doi: 10.1186/s12916-016-0680-9. PMID 27609178
- [Result] Youngster I, Russell GH, Pindar C, Ziv-Baran T, Sauk J, Hohmann EL. Oral, capsulized, frozen fecal microbiota transplantation for relapsing Clostridium difficile infection. JAMA. 2014 Nov 5;312(17):1772-8. doi: 10.1001/jama.2014.13875. PMID 25322359
- [Result] Nash AK, Auchtung TA, Wong MC, Smith DP, Gesell JR, Ross MC, Stewart CJ, Metcalf GA, Muzny DM, Gibbs RA, Ajami NJ, Petrosino JF. The gut mycobiome of the Human Microbiome Project healthy cohort. Microbiome. 2017 Nov 25;5(1):153. doi: 10.1186/s40168-017-0373-4. PMID 29178920
- [Result] Quince C, Walker AW, Simpson JT, Loman NJ, Segata N. Shotgun metagenomics, from sampling to analysis. Nat Biotechnol. 2017 Sep 12;35(9):833-844. doi: 10.1038/nbt.3935. PMID 28898207
- [Result] Langmead B, Salzberg SL. Fast gapped-read alignment with Bowtie 2. Nat Methods. 2012 Mar 4;9(4):357-9. doi: 10.1038/nmeth.1923. PMID 22388286
- [Result] Kao D, Roach B, Silva M, Beck P, Rioux K, Kaplan GG, Chang HJ, Coward S, Goodman KJ, Xu H, Madsen K, Mason A, Wong GK, Jovel J, Patterson J, Louie T. Effect of Oral Capsule- vs Colonoscopy-Delivered Fecal Microbiota Transplantation on Recurrent Clostridium difficile Infection: A Randomized Clinical Trial. JAMA. 2017 Nov 28;318(20):1985-1993. doi: 10.1001/jama.2017.17077. PMID 29183074
- [Result] Beghini F, McIver LJ, Blanco-Miguez A, Dubois L, Asnicar F, Maharjan S, Mailyan A, Manghi P, Scholz M, Thomas AM, Valles-Colomer M, Weingart G, Zhang Y, Zolfo M, Huttenhower C, Franzosa EA, Segata N. Integrating taxonomic, functional, and strain-level profiling of diverse microbial communities with bioBakery 3. Elife. 2021 May 4;10:e65088. doi: 10.7554/eLife.65088. PMID 33944776
- [Result] Vernocchi P, Marini F, Capuani G, Tomassini A, Conta G, Del Chierico F, Malattia C, De Benedetti F, Martini A, Dallapiccola B, van Dijkhuizen EHP, Miccheli A, Putignani L. Fused Omics Data Models Reveal Gut Microbiome Signatures Specific of Inactive Stage of Juvenile Idiopathic Arthritis in Pediatric Patients. Microorganisms. 2020 Oct 6;8(10):1540. doi: 10.3390/microorganisms8101540. PMID 33036309
- [Result] Zhang X, Li L, Mayne J, Ning Z, Stintzi A, Figeys D. Assessing the impact of protein extraction methods for human gut metaproteomics. J Proteomics. 2018 May 30;180:120-127. doi: 10.1016/j.jprot.2017.07.001. Epub 2017 Jul 10. PMID 28705725
- [Result] Distler U, Kuharev J, Navarro P, Tenzer S. Label-free quantification in ion mobility-enhanced data-independent acquisition proteomics. Nat Protoc. 2016 Apr;11(4):795-812. doi: 10.1038/nprot.2016.042. Epub 2016 Mar 24. PMID 27010757
- [Result] Marzano V, Pane S, Foglietta G, Levi Mortera S, Vernocchi P, Onetti Muda A, Putignani L. Mass Spectrometry Based-Proteomic Analysis of Anisakis spp.: A Preliminary Study towards a New Diagnostic Tool. Genes (Basel). 2020 Jun 24;11(6):693. doi: 10.3390/genes11060693. PMID 32599802
- [Result] Cheng K, Ning Z, Zhang X, Li L, Liao B, Mayne J, Stintzi A, Figeys D. MetaLab: an automated pipeline for metaproteomic data analysis. Microbiome. 2017 Dec 2;5(1):157. doi: 10.1186/s40168-017-0375-2. PMID 29197424
- [Result] Alonso-Betanzos A, Bolon-Canedo V. Big-Data Analysis, Cluster Analysis, and Machine-Learning Approaches. Adv Exp Med Biol. 2018;1065:607-626. doi: 10.1007/978-3-319-77932-4_37. PMID 30051410